CLINICAL TRIAL: NCT03959085
Title: A Phase 3 Randomized Trial of Inotuzumab Ozogamicin (NSC#: 772518) for Newly Diagnosed High-Risk B-ALL; Risk-Adapted Post-Induction Therapy for High-Risk B-ALL, Mixed Phenotype Acute Leukemia, and Disseminated B-LLy
Brief Title: Inotuzumab Ozogamicin and Post-Induction Chemotherapy in Treating Patients With High-Risk B-ALL, Mixed Phenotype Acute Leukemia, and B-LLy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL1732; NCI-2019-02845 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL1732 (Other: Children's Oncology Group); AALL1732 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: B Acute Lymphoblastic Leukemia; B Lymphoblastic Lymphoma; Central Nervous System Leukemia; Mixed Phenotype Acute Leukemia; Testicular Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — Specimen Handling; Biopsy; calaspargase pegol; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Inotuzumab Ozogamicin; Leucovorin; Magnetic Resonance Spectroscopy; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisolone; Methylprednisolone; Radiotherapy; Radiation; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm I (HR-FAV B-ALL) (Experimental): See detailed description for Arm I
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Other: Questionnaire Administration; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm II (HR B-ALL CONTROL) (Active Comparator): See detailed description for Arm II.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm III (HR B-ALL EXPERIMENTAL) (Experimental): See detailed description for Arm III.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Biological: Inotuzumab Ozogamicin; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm IV (MPAL) (Experimental): See detailed description for Arm IV.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisolone; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- ARM V (B-LLY) (Experimental): See detailed description for Arm V.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Prednisolone; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
  Arms: ARM V (B-LLY)
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
  Arms: ARM V (B-LLY)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IV, IT, or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC 544; CMC-544; CMC544; Way 207294; WAY-207294
  Arms: Arm III (HR B-ALL EXPERIMENTAL)
Drug: Leucovorin Calcium — Given PO or IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: ARM V (B-LLY)
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Arm I (HR-FAV B-ALL); Arm II (HR B-ALL CONTROL); Arm III (HR B-ALL EXPERIMENTAL); Arm IV (MPAL)
Drug: Methotrexate — Given IT or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IV or IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: ARM V (B-LLY)
Drug: Prednisolone — Given PO or IV
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
  Arms: ARM V (B-LLY); Arm I (HR-FAV B-ALL); Arm II (HR B-ALL CONTROL); Arm IV (MPAL)
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo testicular radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: ARM V (B-LLY); Arm IV (MPAL)
Radiation: Radiation Therapy — Undergo cranial radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: ARM V (B-LLY); Arm II (HR B-ALL CONTROL); Arm III (HR B-ALL EXPERIMENTAL); Arm IV (MPAL)
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial studies whether inotuzumab ozogamicin added to post-induction chemotherapy for patients with High-Risk B-cell Acute Lymphoblastic Leukemia (B-ALL) improves outcomes. This trial also studies the outcomes of patients with mixed phenotype acute leukemia (MPAL), and B-lymphoblastic lymphoma (B-LLy) when treated with ALL therapy without inotuzumab ozogamicin. Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a type of chemotherapy called calicheamicin. Inotuzumab attaches to cancer cells in a targeted way and delivers calicheamicin to kill them. Other drugs used in the chemotherapy regimen, such as cyclophosphamide, cytarabine, dexamethasone, doxorubicin, daunorubicin, methotrexate, leucovorin, mercaptopurine, prednisone, thioguanine, vincristine, and pegaspargase or calaspargase pegol work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This trial will also study the outcomes of patients with mixed phenotype acute leukemia (MPAL) and disseminated B lymphoblastic lymphoma (B-LLy) when treated with high-risk ALL chemotherapy.

The overall goal of this study is to understand if adding inotuzumab ozogamicin to standard of care chemotherapy maintains or improves outcomes in High Risk B-cell Acute Lymphoblastic Leukemia (HR B-ALL). The first part of the study includes the first two phases of therapy: Induction and Consolidation. This part will collect information on the leukemia, as well as the effects of the initial treatment, to classify patients into post-consolidation treatment groups. On the second part of this study, patients with HR B-ALL will receive the remainder of the chemotherapy cycles (interim maintenance I, delayed intensification, interim maintenance II, maintenance), with some patients randomized to receive inotuzumab. The patients that receive inotuzumab will not receive part of delayed intensification. Other aims of this study include investigating whether treating both males and females with the same duration of chemotherapy maintains outcomes for males who have previously been treated for an additional year compared to girls, as well as to evaluate the best ways to help patients adhere to oral chemotherapy regimens. Finally, this study will be the first to track the outcomes of subjects with disseminated B-cell Lymphoblastic Leukemia (B-LLy) or Mixed Phenotype Acute Leukemia (MPAL) when treated with B-ALL chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare in a randomized manner the 5-year disease-free survival (DFS) for children and young adults with High Risk (HR) B-cell acute lymphoblastic leukemia (B-ALL) treated with modified Berlin-Frankfurt-Munster (mBFM) chemotherapy without delayed intensification (DI) part 2, but with the addition of two blocks of inotuzumab ozogamicin, versus those treated with full mBFM chemotherapy backbone including DI Part 2 without the addition of inotuzumab ozogamicin.

SECONDARY OBJECTIVES:

I. To describe the 5-year DFS for a favorable risk subset of National Cancer Institute (NCI) HR B-ALL (HR-Fav) when treated with mBFM chemotherapy with a single high-dose methotrexate (HD-MTX) interim maintenance (IM) phase and treatment duration of 2 years from the start of IM regardless of sex.

II. To determine the toxicity and tolerability of inotuzumab ozogamicin integrated into the mBFM chemotherapy backbone in HR B-ALL including toxicity experienced during phases of therapy subsequent to inotuzumab ozogamicin.

III. To describe the 5-year event-free survival (EFS) for patients with mixed phenotype acute leukemia (MPAL) receiving mBFM HR B-ALL therapy that includes a second IM phase with Capizzi intravenous (IV) methotrexate without leucovorin rescue plus pegaspargase or calaspargase pegol (C-MTX).

IV. To describe the 5-year EFS for patients with disseminated (Murphy stage III-IV) B-cell lymphoblastic lymphoma (B-LLy) receiving mBFM HR B-ALL therapy that includes a second IM phase with C-MTX.

EXPLORATORY OBJECTIVES:

I. To describe the therapy administered, disease response, and survival outcomes of patients with MPAL who come off protocol therapy due to poor disease response to ALL therapy either during Induction, at end of induction (EOI), or at end of consolidation (EOC).

II. To define the prevalence and significance of minimal marrow disease (MMD) at diagnosis and bone marrow minimal residual disease (MRD) at EOI in disseminated B-LLy.

III. To determine the impact of proposed adherence-enhancing interventions on adherence to oral 6-mercaptopurine in patients with ALL.

OUTLINE: All patients receive the same Induction and Consolidation chemotherapy. Patients with HR-Fav B-ALL are assigned to Arm I. Patients with HR B-ALL are randomized to Arm II or III. Patients with MPAL are assigned to Arm IV, and patients with B-LLy are assigned to Arm V.

All patients with B-ALL receive Induction and Consolidation therapy:

INDUCTION: Patients receive cytarabine intrathecally (IT) on day 1 and central nervous system (CNS)2 patients also receive cytarabine IT on days 4, 5 or 6 and 11 or 12. Patients also receive vincristine intravenously (IV) on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes days 1, 8, 15, and 22, pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase intramuscularly (IM) on day 4, and methotrexate IT on days 8 and 29 (and on days 15 and 22 for CNS3 patients). Patients < 10 years old receive dexamethasone orally (PO) twice daily (BID) or IV on days 1-14; patients >= 10 years old receive prednis(ol)one PO BID or IV on days 1-28. Treatment continues for 5 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO once daily (QD) on days 1-14 and 29-42, and methotrexate IT on days 1, 8, 15, and 22 (CNS3 patients receive methotrexate IT on days 1 and 8). Patients also receive vincristine IV on days 15, 22, 43, and 50, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on days 15 and 43. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients with testicular disease at diagnosis that does not resolve by the end of induction will undergo radiation therapy over 12 once daily fractions. Calaspargase pegol can only be given to patients less than 22 years of age.

POST-CONSOLIDATION THERAPY: After Consolidation, based on clinical features and response, patients with B-ALL are designated as HR-Fav or HR B-ALL. Patients with HR-Fav B-ALL are assigned to Arm I. Patients with HR B-ALL are randomized to Arm II or III. Patients with MPAL and B-LLy are assigned to therapy arms (Arms IV and V) that are identical to Arm II. Patients that are < 10 years, have CNS1, no testicular leukemia, with favorable cytogenetics (ETV6 RUNX1 fusion or double trisomies [4 and 10]), =< 24 hours of steroids in the two weeks prior to diagnosis, and EOI MRD < 0.01% are assigned to Arm I. Patients with HR B-ALL who are surface CD22 positive at diagnosis and have MRD < 0.01% by the end of Consolidation, are randomized to either Arm II or III.

ARM I: HR-FAV B-ALL (Patients that are < 10 years, have CNS1 status, no testicular leukemia, with favorable cytogenetics (ETV6 RUNX1 fusion or double trisomies [4 and 10]), =< 24 hours of steroids in the two weeks prior to diagnosis, and EOI MRD < 0.01%)

INTERIM MAINTENANCE: Patients receive vincristine IV on days 1, 15, 29, and 43, high dose methotrexate IV over 24 hours on days 1, 15, 29, and 43, leucovorin PO or IV on days 3-4, 17-18, 31-32, and 45-46, mercaptopurine PO QD on days 1-14, 15-28, 29-42, and 43-56, and methotrexate IT on days 1 and 29. Treatment continues for 9 weeks in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION (PART I): Patients receive methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine IV on days 1, 8, and 15, doxorubicin IV over 1-15 minutes or up to 1 hour on days 1, 8, and 15, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 4. Treatment (Parts I and II of Delayed Intensification) continues for 9 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

DELAYED INTENSIFICATION (PART II): Patients receive cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39, methotrexate IT on days 29 and 36, vincristine IV on days 43 and 50, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 43. Treatment (Parts I and II of Delayed Intensification) continues for 9 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

MAINTENANCE: Patients receive methotrexate IT on days 1 and 29 for cycles 1-4, and day 1 for subsequent cycles. Patients also receive vincristine IV on day 1, prednisolone PO BID or IV on days 1-5, mercaptopurine PO QD on days 1-84, and methotrexate PO on days 8, 15, 22, 29 (excluded in cycles 1-4), 36, 43, 50, 57, 64, 71, and 78. Cycles repeat every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

Patients with HR B-ALL who have MRD < 0.01% by the end of Consolidation, and leukemic blasts positive for surface CD22 at diagnosis are randomized to Arm II or Arm III.

ARM II: HR B-ALL (CONTROL) INTERIM MAINTENANCE I: Patients receive vincristine IV on days 1, 15, 29 and 43, high dose methotrexate IV over 24 hours on days 1, 15, 29 and 43, leucovorin PO or IV on days 3-4, 17-18, 31-32, 45-46, mercaptopurine PO QD on days 1-14, 15-28, 29-42, and 43-56, and methotrexate IT on days 1 and 29. Treatment continues for 9 weeks in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION (PART I): Patients receive methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine IV on days 1, 8, and 15, doxorubicin IV over 1-15 minutes or up to 1 hour on days 1, 8, and 15, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 4. Treatment (Parts I and II of Delayed Intensification) continues for 9 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

DELAYED INTENSIFICATION (PART II): Patients receive cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39, methotrexate IT on days 29 and 36, vincristine IV on days 43 and 50, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 43. Treatment (Parts I and II of Delayed Intensification) continues for 9 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

INTERIM MAINTENANCE II: Patients receive vincristine on days 1, 11, 21, 31 and 41, methotrexate IV over 2-15 minutes or 10-15 minutes on days 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and pegaspargase or calaspargase pegol IV over 1-2 hours on days 2 and 22 (pegaspargase) or 23 (calaspargase) or pegaspargase IM on days 2 and 22. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

ARM III: HR B-ALL (EXPERIMENTAL) INOTUZUMAB OZOGAMICIN (InO) BLOCK 1: Patients receive inotuzumab ozogamicin IV over 60 minutes on days 1, 8, and 15 and methotrexate IT on day 1. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity.

INTERIM MAINTENANCE I: Patients receive vincristine IV on days 1, 15, 29 and 43, high dose methotrexate IV over 24 hours on days 1, 15, 29, and 43, leucovorin PO or IV on days 3-4, 17-18, 31-32, and 45-46, mercaptopurine PO on days 1-14, 15-28, 29-42, and 43-56, and methotrexate IT on days 1 and 29. Treatment continues for 9 weeks in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION (Part I): Patients receive methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine IV on days 1, 8, and 15, doxorubicin IV over 1-15 minutes or up to 1 hour on days 1, 8, and 15, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 4. Treatment (Parts I and II of Delayed Intensification) continues for 5 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

InO BLOCK 2: Patients receive inotuzumab ozogamicin IV over 60 minutes on days 1, 8, and 15. Treatment continues for 4 weeks in the absence of disease progression or unacceptable toxicity.

INTERIM MAINTENANCE II: Patients receive vincristine IV on days 1, 11, 21, 31, and 41, methotrexate IV on days 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and pegaspargase or calaspargase pegol IV over 1-2 hours on days 2 and 22 (pegaspargase) or 23 (calaspargase) or pegaspargase IM on days 2 and 22. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

ARMS II AND III: HR B-ALL MAINTENANCE: Patients receive vincristine IV on day 1, prednisolone PO BID or IV on days 1-5, mercaptopurine PO on days 1-84, methotrexate PO on days 8, 15, 22, 29 (excluded in cycles 1 and 2), 36, 43, 50, 57, 64, 71 and 78, and methotrexate IT on days 1 (and 29 of cycles 1-2 for patients who do not receive cranial radiation). Cycles repeat every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients with CNS3 disease undergo cranial radiation therapy over 10 fractions during the first 4 weeks.

ARM IV: MPAL INDUCTION: Patients receive cytarabine IT on day 1 and CNS2 patients also receive cytarabine IT on days 4, 5 or 6 and 11 or 12. Patients also receive vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes days 1, 8, 15, and 22, pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 4, and methotrexate IT on days 8 and 29 (and on days 15 and 22 for CNS3 patients). Patients < 10 years old receive dexamethasone PO BID or IV on days 1-14; patients >= 10 years old receive prednisolone PO BID or IV on days 1-28. Treatment continues for 5 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine IV over 1-30 minutes or SC on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO on days 1-14 and 29-42, methotrexate IT on days 1, 8, 15, and 22 (excluded on days 15 and 22 for CNS3 patients), vincristine IV on days 15, 22, 43, and 50, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on days 15 and 43. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients with testicular disease at diagnosis that does not resolve by the end of induction will and continued evidence of testicular disease at end of induction undergo testicular radiation over 12 once-daily fractions. Calaspargase pegol can only be given to patients less than 22 years of age.

ARM V: B-LLY INDUCTION: Patients receive cytarabine IT on day 1 and CNS2 patients also receive cytarabine IT on days 4, 5 or 6 and 11 or 12. Patients also receive vincristine IV on days 1, 8, 15, and 22, daunorubicin IV over 1-15 minutes days 1, 8, 15, and 22, pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 4, and methotrexate IT on days 8 and 29 (and on days 15 and 22 for CNS3 patients). Patients < 10 years old receive dexamethasone PO BID or IV on days 1-14; patients >= 10 years old receive prednisolone PO BID or IV on days 1-28. Treatment continues for 5 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

CONSOLIDATION: Patients receive cyclophosphamide IV over 30-60 minutes on days 1 and 29, cytarabine IV over 1-30 minutes or SC on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO on days 1-14 and 29-42, methotrexate IT on days 1, 8, 15, and 22 (excluded on days 15 and 22 CNS3 patients), vincristine IV on days 15, 22, 43, and 50, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on days 15 and 43. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients with testicular disease at diagnosis that does not resolve by the end of induction will and continued evidence of testicular disease at end of induction undergo testicular radiation therapy over 12 once-daily fractions. Calaspargase pegol can only be given to patients less than 22 years of age.

ARM IV AND V: MPAL AND B-LLY (Post-Consolidation Therapy) INTERIM MAINTENANCE I: Patients receive vincristine IV on days 1, 15, 29, and 43, high dose methotrexate IV over 24 hours on days 1, 15, 29, and 43, leucovorin PO or IV on days 3-4, 17-18, 31-32, and 45-46, methotrexate IT on days 1 and 29 and mercaptopurine PO QD on days 1-14, 15-28, 29-42, and 43-56. Treatment continues for 9 weeks in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION (PART I): Patients receive methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-7 and 15-21, vincristine IV on days 1, 8, and 15, doxorubicin IV over 1-15 minutes or up to 1 hour on days 1, 8, and 15, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 4. Treatment (Parts I and II of Delayed Intensification) continues for 9 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

DELAYED INTENSIFICATION (PART II): Patients receive cyclophosphamide IV over 30-60 minutes on day 29, thioguanine PO on days 29-42, cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39, methotrexate IT on days 29 and 36, vincristine IV or IV push over 1 minute on days 43 and 50, and pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase IM on day 43. Treatment (Parts I and II of Delayed Intensification) continues for 9 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

INTERIM MAINTENANCE II: Patients receive vincristine IV on days 1, 11, 21, 31, and 41, methotrexate IV or infusion over 2-15 minutes or 10-15 minutes on days 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and pegaspargase or calaspargase pegol IV over 1-2 hours on days 2 and 22 (pegaspargase) or (calaspargase) 23 or pegaspargase IM on days 2 and 22. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Calaspargase pegol can only be given to patients less than 22 years of age.

MAINTENANCE: Patients receive vincristine IV on days 1, prednisolone PO BID or IV on days 1-5, mercaptopurine PO on days 1-84, methotrexate PO on days 8, 15, 22, 29 (excluded in cycles 1 and 2), 36, 43, 50, 57, 64, 71, and 78, and methotrexate IT on days 1 (and 29 of cycles 1-2 for patients who do not receive cranial radiation). Cycles repeat every 12 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients with CNS3 disease at diagnosis undergo cranial radiation therapy for 10 fractions over 4 weeks.

Patients undergo blood sample collection and bone marrow aspiration and biopsy on study. B-LLy patients undergo computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), and/or bone scan on study.

After completion of study treatment, patients are followed up at 4 weeks, then every 3 months for 2 years, every 4-6 months for the third year, then every 6-12 months for years 4-5.

ELIGIBILITY:
Inclusion Criteria:

* B-ALL and MPAL patients must be enrolled on APEC14B1 and consented to eligibility studies (Part A) prior to treatment and enrollment on AALL1732. Note that central confirmation of MPAL diagnosis must occur within 22 days of enrollment for suspected MPAL patients. If not performed within this time frame, patients will be taken off protocol.
* APEC14B1 is not a requirement for B-LLy patients but for institutional compliance every patient should be offered participation in APEC14B1. B-LLy patients may directly enroll on AALL1732.
* Patients must be > 365 days and < 25 years of age
* White blood cell count (WBC) criteria for patients with B-ALL (within 7 days prior to the start of protocol-directed systemic therapy):

  * Age 1-9.99 years: WBC >= 50,000/uL
  * Age 10-24.99 years: Any WBC
  * Age 1-9.99 years: WBC < 50,000/uL with:

    * Testicular leukemia
    * CNS leukemia (CNS3)
    * Steroid pretreatment.
* White blood cell count (WBC) criteria for patients with MPAL (within 7 days prior to the start of protocol-directed systemic therapy):

  * Age 1-24.99 years: any WBC NOTE: Patients enrolled as suspected MPAL but found on central confirmatory testing to have B-ALL must meet the B-ALL criteria above (age, WBC, extramedullary disease, steroid pretreatment) to switch to the B-ALL stratum before the end of induction.
* Patient has newly diagnosed B-ALL or MPAL (by World Health Organization [WHO] 2016 criteria) with >= 25% blasts on a bone marrow (BM) aspirate;

  * OR If a BM aspirate is not obtained or is not diagnostic of acute leukemia, the diagnosis can be established by a pathologic diagnosis of acute leukemia on a BM biopsy;
  * OR A complete blood count (CBC) documenting the presence of at least 1,000/uL circulating leukemic cells if a bone marrow aspirate or biopsy cannot be performed.
* Patient has newly diagnosed B-LLy Murphy stages III or IV.
* Patient has newly diagnosed B-LLy Murphy stages I or II with steroid pretreatment.
* Note: For B-LLy patients with tissue available for flow cytometry, the criterion for diagnosis should be analogous to B-ALL. For tissue processed by other means (i.e., paraffin blocks), the methodology and criteria for immunophenotypic analysis to establish the diagnosis of B-LLy defined by the submitting institution will be accepted.
* Central nervous system (CNS) status must be determined prior to enrollment based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment and cytoreduction. It is recommended that intrathecal cytarabine be administered at the time of the diagnostic lumbar puncture. This is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture. This is allowed prior to enrollment. Systemic chemotherapy must begin within 72 hours of this intrathecal therapy.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and NCI requirements for human studies must be met.

Exclusion Criteria:

* Patients with Down syndrome are not eligible (patients with Down syndrome and B-ALL are eligible for AALL1731, regardless of NCI risk group).
* With the exception of steroid pretreatment and steroid cytoreduction or the administration of intrathecal cytarabine, patients must not have received any prior cytotoxic chemotherapy for the current diagnosis of B-ALL, MPAL, or B-LLy or for any cancer diagnosed prior to initiation of protocol therapy on AALL1732.
* Patients who have received > 72 hours of hydroxyurea within one week prior to start of systemic protocol therapy.
* Patients with B-ALL or MPAL who do not have sufficient diagnostic bone marrow submitted for APEC14B1 testing and who do not have a peripheral blood sample submitted containing > 1,000/uL circulating leukemia cells.
* Patients with acute undifferentiated leukemia (AUL) are not eligible.
* For Murphy stage III/IV B-LLy patients, or stage I/II patients with steroid pretreatment, the following additional exclusion criteria apply:

  * T-lymphoblastic lymphoma.
  * Morphologically unclassifiable lymphoma.
  * Absence of both B-cell and T-cell phenotype markers in a case submitted as lymphoblastic lymphoma.
* Patients with known Charcot-Marie-Tooth disease.
* Patients with known MYC translocation associated with mature (Burkitt) B-cell ALL, regardless of blast immunophenotype.
* Patients requiring radiation at diagnosis.
* Female patients who are pregnant, since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.
* Lactating women who plan to breastfeed their infants while on study and for 2 months after the last dose of inotuzumab ozogamicin.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of study participation. For those patients randomized to inotuzumab ozogamicin, there is a minimum of 8 months after the last dose of inotuzumab ozogamicin for females and 5 months after the last dose of inotuzumab ozogamicin for males.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4997 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in 5-year disease-free survival (DFS) | From end of consolidation (EOC) to first event (relapse, second malignant neoplasm, remission death) or date of last contact, assessed up to 5 years
  Improvement in 5-year disease-free survival (DFS) with modified Berlin-Frankfurt-Münster (mBFM) chemotherapy without delayed intensification (DI) part 2 but with inotuzumab ozogamicin, versus full mBFM chemotherapy backbone including DI Part 2 without the addition of inotuzumab ozogamicin. Power calculations are based on detecting an improvement in post consolidation DFS with the addition of InO to standard therapy for high risk (HR) B-acute lymphoblastic leukemia (ALL). All survival time analyses assume a Weibull distribution with shape parameter of 0.6 (based on historical data). Will be estimated using the Kaplan-Meier method and standard errors and confidence intervals estimated by the method of Peto. Estimation of treatment effect will be done using intent-to-treat (ITT) analysis based on randomized group.

SECONDARY OUTCOMES:
5-year DFS for favorable risk subset of NCI HR B-ALL (HR favorable) when treated with mBFM chemotherapy with a single high-dose methotrexate (HD MTX) Interim Maintenance (IM) phase and treatment duration of 2 years from the start of IM regardless of sex | From EOC to first event (relapse, second malignant neoplasm, remission death) or date of last contact, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method and standard errors and confidence intervals estimated by the method of Peto. Estimation of treatment effect will be done using ITT analysis based on randomized group.
Incidence of adverse events for the integration of inotuzumab ozogamicin into the mBFM chemotherapy backbone in HR B-ALL | Up to 5 years
  Graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will be monitored and reported.
5-year event-free survival (EFS) for patients with mixed phenotype acute leukemia (MPAL) receiving mBFM HR B-ALL therapy that includes a second IM phase with Capizzi escalating intravenous MTX without leucovorin rescue + pegaspargase or calapargase pegol | From study entry to first event (induction failure, Induction death, end of induction (EOI) minimal residual disease (MRD) >= 5%, EOC MRD >= 0.01%, relapse, second malignancy, remission death) or date of last contact, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method and standard errors and confidence intervals estimated by the method of Peto. Estimation of treatment effect will be done using ITT analysis based on randomized group.
5-year EFS for patients with disseminated (Murphy stage III-IV) B-cell lymphoblastic lymphoma (B-LLy) receiving mBFM HR B-ALL therapy that includes a second IM phase with C-MTX | From study entry to first event (progressive disease, induction death, relapse, second malignancy, remission death) or date of last contact, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method and standard errors and confidence intervals estimated by the method of Peto. Estimation of treatment effect will be done using ITT analysis based on randomized group.
Overall survival (OS) | Time from study entry to death or date of last contact for those alive at last contact, assessed up to 5 years
  OS rates will be estimated using the Kaplan-Meier method and standard errors and confidence intervals estimated by the method of Peto.

OTHER OUTCOMES:
Therapy administered to patients with MPAL who come off protocol therapy due to poor disease response to ALL therapy | Up to 5 years
  Will be described.
Disease response in patients with MPAL who come off protocol therapy due to poor disease response to ALL therapy | Up to 5 years
  Will be described.
Survival outcomes of patients with MPAL who come off protocol therapy due to poor disease response to ALL therapy | Up to 5 years
  Will be described.
Prevalence and significance of minimal marrow disease (MMD) at diagnosis and bone marrow MRD in disseminated B-LLy | Up to 5 years
  Percentages with MMD at induction and MRD positivity at end of Induction will be described.
Impact of four proposed interventions of varying intensities to enhance adherence to oral 6 mercaptopurine, with a randomization based upon baseline adherence measured during the first cycle of maintenance therapy | Up to 5 years
  The main analyses will use mixed models including random effects to account for the multiple sites and longitudinal observations within patients. Will examine unadjusted associations of the primary outcome (MEMS-based adherence rate) with demographic, clinical and sociodemographic variables for the entire cohort (across 3 intervention arms). Those patient-level factors associated with the outcome will be included in the main model as fixed effects to improve the precision of the estimates. The basic model for adherence will include time and mean adherence during the baseline pre-intervention period and treatment group. It will also include interactions between time and both baseline adherence and intervention group to allow for intervention-specific trends and normal changes in adherence over time.
DFS by sex | Up to 5 years
  Estimates of DFS and the corresponding 95% confidence intervals by sex.
DFS by race | Up to 5 years
  Estimates of DFS and the corresponding 95% confidence intervals by race.
DFS by ethnicity | Up to 5 years
  Estimates of DFS and the corresponding 95% confidence intervals by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L McNeer, Principal Investigator — Children's Oncology Group
Locations (230):
- United States (203):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Vannie Cook Children's Clinic, McAllen, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - University Pediatric Hospital, San Juan